CLINICAL TRIAL: NCT02973945
Title: High Flow Nasal Cannula Versus The Venturi Mask During Exercise Training in Chronic Obstructive Pulmonary Disease Patients, a Randomized, Simple Blind, Controlled Trial.
Brief Title: High Flow Nasal Cannula and Aerobic Capacity Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3011
Record Dates: First submitted 2016-11-10; First posted 2016-11-28 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-05

CONDITIONS: COPD
Keywords: Pulmonary Rehabilitation; High Flow Nasal Cannula; The Venturi Mask; Exercise capacity; Aerobic capacity; HFNC
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (Experimental): During a 8 week Pulmonary Rehabilitation Program patients will receive oxygen through High Flow Nasal Cannula (HFNC) while they are training aerobic capacity on the treadmill.
  Interventions: Device: High Flow Nasal Cannula
- The Venturi Mask (Active Comparator): During a 8 week Pulmonary Rehabilitation Program patients will receive oxygen through The Venturi Mask (VM) while they are training aerobic capacity on the treadmill.
  Interventions: Device: The Venturi Mask

INTERVENTIONS:
Device: High Flow Nasal Cannula — During the pulmonary rehabilitation program, patients will train the aerobic capacity on a treadmill. Patients in the intervention arm will receive oxygen trough High Flow Nasal Cannula (HFNC) at 50 lpm and 40% of oxygen.
  The aerobic capacity training plan will be conducted three times a week over 24 sessions.
  Other Names: HFNC
  Arms: High Flow Nasal Cannula
Device: The Venturi Mask — During the pulmonary rehabilitation program, patients will train the aerobic capacity on a treadmill. Patients in the control arm will receive oxygen trough The Venturi Mask (VM) at 40% of oxygen.
  The aerobic capacity training plan will be conducted three times a week over 24 sessions.
  Other Names: VM
  Arms: The Venturi Mask

SUMMARY:
The aim of this study is to compare exercise capacity in Chronic Obstructive Pulmonary Disease (COPD) patients before and after an 8 week pulmonary rehabilitation program.

Patients will be randomised in two groups, one arm will received oxygen through High Flow Nasal Cannula (HFNC) and the other group by The Venturi Mask (VM)

DETAILED DESCRIPTION:
Design: randomized, single blind, controlled trial.

The main goal of this study is to compare the exercise tolerance in COPD patients after an 8 week pulmonary rehabilitation program using High Flow Nasal Cannula or The Venturi Mask. The exercise tolerance will be measured in seconds in a Constant Load Treadmill Test (CTLT).

ELIGIBILITY:
Inclusion Criteria:

1. Long term oxygen therapy (LTOT) or oxygen needs during exercise.
2. Clinically stable defined as four weeks without exacerbation

Exclusion Criteria:

1. Refusal to participate
2. Any neuromuscular, cardiovascular or any other condition that limits test performance.
3. Contraindication for exercise

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Capacity - Maximum Walking Time Reached | 8 weeks
  The exercise capacity test measures the maximum time (in minutes) reached during a Constant Load Treadmill Test (CLTT).
  The treadmill speed will be constant and set up at 90% of the maximum speed reached in the previous Incremental Load Treadmill Test (ILTT).
  The patient will walk at the same velocity until he exhausts his capacity thus ending the test.
  This CLTT will be performed three times, always after an Incremental Load Treadmill Test (ILTT)

SECONDARY OUTCOMES:
Six Minutes Walking Test | 8 weeks
  A Six Minute Walking Test will be conducted according to American Thoracic Society (ATS) guide.
  Patients will be asked to walk as much as they can in that period of time. During the test oxygen saturation and cardiac frequency will be recorded.
Exercise capacity - Maximum Walking Speed Reached | 8 weeks
  The exercise capacity test measures the maximum speed (in Km/h) reached during an Incremental Load Treadmill Test (ILTT).
  The test begins at a speed of 3km/h and each minute after will increase by 0.5 km/h.
  The patient will walk until he exhausts his capacity, once reached, the test will finished.
  This ILTT will be performed three times, always before the Constant Load Treadmill Test (CLTT)
Quality of Life - The St George's Respiratory Questionnaire | 8 weeks
  The St George's Respiratory Questionnaire (SGRQ) is an instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.
Quality of Life -Chronic Obstructive Pulmonary Disease Assessment Test | 8 weeks
  The Chronic Obstructive Pulmonary Disease Assessment Test (CAT) is a patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dyspnea, chest tightness) on health status.
Dyspnea | 8 weeks
  The modified Medical research Council Scale (0-4) will be used in order to assess the breathless subjective sensation.
Comfort | 8 weeks
  Difference in global comfort according to the device used with visual analogue scale (VAS) 0-10 between High Flow Nasal Cannula and The Venturi Mask

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas NR Roux, PT-RT, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos AIres, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Rabinovich RA, Vilaro J. Structural and functional changes of peripheral muscles in chronic obstructive pulmonary disease patients. Curr Opin Pulm Med. 2010 Mar;16(2):123-33. doi: 10.1097/MCP.0b013e328336438d. PMID 20071991
- [Result] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Result] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Result] Guell Rous MR, Diaz Lobato S, Rodriguez Trigo G, Morante Velez F, San Miguel M, Cejudo P, Ortega Ruiz F, Munoz A, Galdiz Iturri JB, Garcia A, Servera E; Sociedad Espanola de Neumologia y Cirugia Toracica (SEPAR). Pulmonary rehabilitation. Sociedad Espanola de Neumologia y Cirugia Toracica (SEPAR). Arch Bronconeumol. 2014 Aug;50(8):332-44. doi: 10.1016/j.arbres.2014.02.014. Epub 2014 May 17. English, Spanish. PMID 24845559
- [Result] Sivori M, Almeida M, Benzo R, Boim C, Brassesco M, Callejas O, Capparelli I, Conti E, Diaz M, Draghi J, Franco J, Gando S, Giuliano G, Guida R, Jolly E, Pessolano F, Rabinovich R, Ratto P, Rhodius E, Saadia M, Salvado A, Sobrino E, Victorio C. [New argentine consensus of respiratory rehabilitation 2008]. Medicina (B Aires). 2008;68(4):325-44. Spanish. PMID 18786894
- [Result] O'Donnell DE, D'Arsigny C, Webb KA. Effects of hyperoxia on ventilatory limitation during exercise in advanced chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Mar;163(4):892-8. doi: 10.1164/ajrccm.163.4.2007026. PMID 11282762
- [Result] Maltais F, Simon M, Jobin J, Desmeules M, Sullivan MJ, Belanger M, Leblanc P. Effects of oxygen on lower limb blood flow and O2 uptake during exercise in COPD. Med Sci Sports Exerc. 2001 Jun;33(6):916-22. doi: 10.1097/00005768-200106000-00010. PMID 11404656
- [Result] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Result] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Result] Cirio S, Piran M, Vitacca M, Piaggi G, Ceriana P, Prazzoli M, Paneroni M, Carlucci A. Effects of heated and humidified high flow gases during high-intensity constant-load exercise on severe COPD patients with ventilatory limitation. Respir Med. 2016 Sep;118:128-132. doi: 10.1016/j.rmed.2016.08.004. Epub 2016 Aug 8. PMID 27578482
- [Result] Hardinge M, Suntharalingam J, Wilkinson T; British Thoracic Society. Guideline update: The British Thoracic Society Guidelines on home oxygen use in adults. Thorax. 2015 Jun;70(6):589-91. doi: 10.1136/thoraxjnl-2015-206918. Epub 2015 Apr 27. PMID 25918120
- [Result] Puente-Maestu L, Palange P, Casaburi R, Laveneziana P, Maltais F, Neder JA, O'Donnell DE, Onorati P, Porszasz J, Rabinovich R, Rossiter HB, Singh S, Troosters T, Ward S. Use of exercise testing in the evaluation of interventional efficacy: an official ERS statement. Eur Respir J. 2016 Feb;47(2):429-60. doi: 10.1183/13993003.00745-2015. Epub 2016 Jan 21. PMID 26797036
- [Result] Cooper CB, Abrazado M, Legg D, Kesten S. Development and implementation of treadmill exercise testing protocols in COPD. Int J Chron Obstruct Pulmon Dis. 2010 Oct 12;5:375-85. doi: 10.2147/copd.s11153. PMID 21103404
- [Result] Marrugat J, Vila J, Pavesi M, Sanz F. [Estimation of the sample size in clinical and epidemiological investigations]. Med Clin (Barc). 1998 Sep 12;111(7):267-76. No abstract available. Spanish. PMID 9789243
- [Result] ERS Task Force; Palange P, Ward SA, Carlsen KH, Casaburi R, Gallagher CG, Gosselink R, O'Donnell DE, Puente-Maestu L, Schols AM, Singh S, Whipp BJ. Recommendations on the use of exercise testing in clinical practice. Eur Respir J. 2007 Jan;29(1):185-209. doi: 10.1183/09031936.00046906. PMID 17197484
- [Result] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Result] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Result] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Result] Laszlo G. Standardisation of lung function testing: helpful guidance from the ATS/ERS Task Force. Thorax. 2006 Sep;61(9):744-6. doi: 10.1136/thx.2006.061648. PMID 16936234
- See also: Global initiative for Chronic Obstructive Lung Disease. Update 2016 — http://goldcopd.org/